CLINICAL TRIAL: NCT01651689
Title: Hair Counts From Vertical and Horizontal Sections of Scalp Biopsy SPecimens in Thai Population With Alopecia
Acronym: ThaiScalpBx
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Assistant Professor, Siriraj Hospital
Other Study IDs: SirirajH-003; 553/2553(EC3) (Registry Identifier: 553/2553(EC3))
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Alopecia
Keywords: Scalp biopsy; Hair count; Vertical section; Horizontal section; Thais
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — scalp biopsy specimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Scalp biopsy: Subjects are on scadule list for hair transplantation in Siriraj hospital. Scalp biopsy with punch biopsy No.4 Scalp biopsy by punch biopsy No.4 at occipital area was done in subjects who have hair transplantaion.

SUMMARY:
Hair disorders, expecialy scarring alopecia were diagnosed by scalp biopsy specimens in horizontal and vertical sections.(1-4) Data on hair density in Thais are lacking, although in Asians have more fewer hairs than whites.(5-7)Howevery, previous study from East Asian just had only one study and the data was more differently from West Asian and whites. Then this study was performed to evaluate hair density in Thais, and compared to previous study.

ELIGIBILITY:
Inclusion Criteria:

* Thai
* Age >= 18 years
* Diagnosis alopecia and on list for hair transplantation in Siriraj hospital

Exclusion Criteria:

* Alopecia areata or positive hair pulling test
* Underlying disease : DM, chronic renal failure, chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai patients who have alopecia and on scadule for hair transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rattapon Thuangtong, MD, Principal Investigator — Department of Dermatology, Siriraj hospital, Faculty of Medicine, Mahidol University, Thailand
Locations (1):
- Siriraj hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Elston DM, McCollough ML, Angeloni VL. Vertical and transverse sections of alopecia biopsy specimens: combining the two to maximize diagnostic yield. J Am Acad Dermatol. 1995 Mar;32(3):454-7. doi: 10.1016/0190-9622(95)90068-3. PMID 7868715
- [Background] Elston DM, Ferringer T, Dalton S, Fillman E, Tyler W. A comparison of vertical versus transverse sections in the evaluation of alopecia biopsy specimens. J Am Acad Dermatol. 2005 Aug;53(2):267-72. doi: 10.1016/j.jaad.2005.03.007. PMID 16021122
- [Background] Garcia C, Poletti E. Scalp biopsy specimens: transverse vs vertical sections. Arch Dermatol. 2007 Feb;143(2):268. doi: 10.1001/archderm.143.2.268-a. No abstract available. PMID 17310014
- [Background] Elston DM. Vertical vs. transverse sections: both are valuable in the evaluation of alopecia. Am J Dermatopathol. 2005 Aug;27(4):353-6. doi: 10.1097/01.dad.0000164602.10908.92. No abstract available. PMID 16121061
- [Background] Sperling LC. Hair density in African Americans. Arch Dermatol. 1999 Jun;135(6):656-8. doi: 10.1001/archderm.135.6.656. PMID 10376692
- [Background] Lee HJ, Ha SJ, Lee JH, Kim JW, Kim HO, Whiting DA. Hair counts from scalp biopsy specimens in Asians. J Am Acad Dermatol. 2002 Feb;46(2):218-21. doi: 10.1067/mjd.2002.119558. PMID 11807433
- [Background] Aslani FS, Dastgheib L, Banihashemi BM. Hair counts in scalp biopsy of males and females with androgenetic alopecia compared with normal subjects. J Cutan Pathol. 2009 Jul;36(7):734-9. doi: 10.1111/j.1600-0560.2008.01149.x. PMID 19519605